CLINICAL TRIAL: NCT04392401
Title: Study of the Kinetics of the Immune Response During the Intensive Care Unit Stay in Adult Patients Infected With SARS-CoV-2: Multicentric Non Interventional Study
Brief Title: COVID-19 - Study of the Kinetics of the Immune Response During the Intensive Care Unit Stay in Adult Patients Infected With SARS-CoV-2: Multicentric Non Interventional Study
Acronym: RICO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0358; 2020-A01079-30 (Other: ANSM)
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Intensive Care Unit; SARS-Cov-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — one EDTA sample and one PAXGENETM sample will be collected at Day 0, Day 3, Day 7, Day 12 and Day 20 in order to analyze immune system response
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients over 18 years with a confirmed diagnosis of COVID 19 hospitalized in intensive care unit
  Interventions: Biological: Collection of blood samples in order to create a biocollection

INTERVENTIONS:
Biological: Collection of blood samples in order to create a biocollection — Blood samples will be collected at admission in intensive care, at Day 3, Day 7, Day 12 and Day 20 during their hospitalization. Clinical data from routine care will be collected. Vital status will be assessed at Day 28 and Day 90.

SUMMARY:
Infection with the SARS-CoV-2 coronavirus (COVID-19) has recently been identified as a pandemic due to the speed and global scale of its transmission. In Auvergne-Rhône-Alpes region (AURA), the epidemic began in February 2020 and the number of infected people is still important. Between 15 and 20% of COVID-19 patients develop an acute respiratory distress syndrome (ARDS) leading to their hospitalization in intensive care. Their clinical progression can be rapidly harmful with the development of severe ARDS associated with an increased risk of death.

Preliminary data on the immune response of COVID-19 patients describe the induction of a moderate inflammatory response and the occurrence of major progressive lymphopenia over time associated with potential immunosuppression. Up to 50% of secondary infections are reported in deceased COVID-19 patients. However, no prospective study has exhaustively described the kinetics of the immune response of COVID-19 patients in intensive care.

The precise description of the immune response over time in adult patients with a proven infection with the SARS-CoV-2 virus and the study of the relation between this response and the increased risk of organ failure (severe ARDS), death or nosocomial infection will allow us to better understand the pathophysiology of the immune response induced by COVID-19 in order to (i) identify new therapeutic strategies targeting the host response in patients in intensive care (ii) to develop biological markers to stratify patients for future clinical trials evaluating these immunoadjuvant treatments in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged 18 or over,
2. Hospitalization in intensive care for Sars-Cov-2 pneumopathy,
3. First hospitalization in intensive care unit,
4. Positive diagnosis of SARS-CoV2 infection carried out by PCR or by another approved method in at least one respiratory sample,
5. Sampling in the first 24 hours after admission to intensive care unit (D0 / D1) feasible,
6. Patient or next of kin who has been informed of the terms of the study and has not objected to participating.

Exclusion Criteria:

1. Pregnant or lactating woman,
2. Person placed under legal protection,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in intensive care unit for the management of a SARS-CoV-2 pulmonary infection confirmed by PCR diagnosis or according to the approved method at the time of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Kinetics over time of HLA-DR expression on the surface of monocytes | Along the intensive care stay, an average of 20 days
  Kinetics along the intensive care stay of HLA-DR expression on the surface of monocytes expressed as the number of antibodies fixed per cell

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne VENET, Principal Investigator — Hospices Civils de Lyon
Locations (7):
- France (7):
  - Hôpital Pierre Wertheimer, Bron
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre hospitalier universitaire de Grenoble Alpes, Grenoble
  - Hôpital Edouard Herriot, Lyon
  - Hôpial de la Croix Rousse, Lyon
  - Hôpital Lyon Sud, Pierre-Bénite
  - CH de St Etienne, Saint-Etienne

REFERENCES:
- [Derived] Bidar F, Hamada S, Gossez M, Coudereau R, Lopez J, Cazalis MA, Tardiveau C, Brengel-Pesce K, Mommert M, Buisson M, Conti F, Rimmele T, Lukaszewicz AC, Argaud L, Cour M, Monneret G, Venet F; RICO Study Group. Recombinant human interleukin-7 reverses T cell exhaustion ex vivo in critically ill COVID-19 patients. Ann Intensive Care. 2022 Mar 5;12(1):21. doi: 10.1186/s13613-022-00982-1. PMID 35246776